CLINICAL TRIAL: NCT04297436
Title: Use of Bexsero Immunisation to Detect Cross Reactive Antigens and Anti-gonococcal Antibodies in Key Populations in Kenya
Brief Title: Gonococcal Vaccine Study in Key Populations in Kenya
Acronym: BexKPK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: KEMRI-Wellcome Trust Collaborative Research Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CSC 182; OXTREC16-20 (Other: University of Oxford)
Record Dates: First submitted 2020-02-27; First posted 2020-03-05 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Gonorrhea
MeSH Terms: conditions — Gonorrhea | interventions — 4CMenB vaccine; Vaccines

STUDY DESIGN:
Intervention Model Description: To assess if immunisation of individuals at risk for gonococcal infection with 4CMenB (Bexsero) elicits humoral and T cell cross-reactive responses against Neisseria gonorrhoeae (Ng)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bexsero (Other): Each participant is compared to baseline (before vaccination)
  Interventions: Biological: 4CMenB (Bexsero®) vaccine

INTERVENTIONS:
Biological: 4CMenB (Bexsero®) vaccine — Tthe 4CMenB vaccine (Bexsero®) contains the MeNZB OMV component plus three recombinant antigens (NadA, fHBP-GNA2091, and NHBA-GNA1030. The 4CMenB vaccine (Bexsero®) induces antibodies in humans that recognise gonococcal proteins.

SUMMARY:
Gonorrhoea is a sexually transmitted infection that can infect both men and women. It can cause infections in the genitals, rectum, and throat. It is a very common infection, especially among young people aged 18-25 years.

Meningococcal disease and gonorrhoea are caused by bacteria that are closely related but cause different diseases that are spread in different ways. New evidence suggests that the Meningococcal B vaccine (Bexsero®) licensed outside of Kenya against meningococcal B disease may also be effective against gonorrhoea due to genetic similarities between the two organisms causing the two diseases. The aim of this study is to generate data to develop a gonorrhoea vaccine, using an existing vaccine against meningococcal disease

DETAILED DESCRIPTION:
Meningococcal disease and gonorrhoea are caused by bacteria that are closely related but cause different diseases that are spread in different ways. New evidence suggests that the Meningococcal B vaccine (Bexsero®) licensed outside of Kenya against meningococcal B disease may also be effective against gonorrhoea due to genetic similarities between the two organisms causing the two diseases. Investigators will conduct a clinical trial of the Meningococcal B vaccine (Bexsero®) in approximately 50 male and female participants aged 18-25 years who are in follow up in KEMRI cohorts (including HIV-uninfected and infected individuals) at the KEMRI clinic in Mtwapa. This is not an efficacy trial. Instead, investigators will assess if immunisation of individuals at risk for gonococcal infection with 4CMenB (Bexsero®) elicits humoral and T cell cross-reactive responses against Neisseria gonorrhoeae (Ng). Participants will make six study visits, including a screening visit, an enrolment visit and 4 follow up visits. InvestigatorsF will offer vaccination with the Meningococcal B vaccine (Bexsero®) vaccine at the enrolment visit and approximately 2 months later. Investigators will collect a 20ml blood sample at enrolment, and following the first vaccination, and a 70ml blood sample following the second vaccination. At study completion (month 6), investigators will collect a 4ml blood sample. Investigators will collect a throat swab, a urine sample (for men), vaginal swab, and an anal swab at the enrolment, month 3 and month 6 visit to test for Chlamydiae and Gonorrhoea infection. Total study participation for participants is 6 months. Upon study completion, participants will continue to receive research care at the KEMRI clinic in Mtwapa.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female as assessed by a medical history, physical exam, and laboratory tests (specified in study operations manual).
* At least 18 years of age on the day of screening and will not reach 26th birthday on the day of the second vaccination (approximately 6 weeks after enrolment)
* Willing and able to give informed consent for participation in the trial before any study-related procedures are performed.
* Willing to donate blood samples for immunogenicity assessments.

Exclusion Criteria:

Any clinically significant acute or chronic medical condition that is considered progressive that, in the opinion of the Principal Investigator or designee, makes the volunteer unsuitable for participation in the trial

* Pregnancy
* Participation in another clinical trial (i.e. investigational HIV vaccine candidate), within the previous 3 months or expected participation during the study
* Bleeding disorder diagnosed by a physician (e.g., factor deficiency, coagulopathy or platelet disorder that requires special precautions).
* History of severe local or systemic reactogenicity to vaccines (e.g., anaphylaxis, respiratory difficulty, angioedema).

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
humoral and T cell cross-reactive responses against Neisseria gonorrhoeae | approximately 2 weeks following completed vaccination (2 doses)
  Serum antigen- and OMV-specific IgG1, IgG2a, Ig3A and IgA titres will be determined.
  T cell responses will be measured in two ways:
  Indirect responses: by determining the IgG1/IgG2 ratios after immunization. Direct responses: PBMCs will be isolated at enrolment, 2 weeks post second immunization and used for the detection of antigen-specific IFN secreting T cells.
  The induction of antibody will be measured by a standard endpoint ELISA assay using peptides covering recombinant protein antigens, purified antigens, and defined OMVs.
  After the final immunization, PBMCs will be collected for isolation of antigen-specific memory B cells, aiming to generate human monoclonal antibodies (mAbs) against key vaccine candidates.

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Sanders, MD, PhD, Principal Investigator — University of Oxford & KEMRI-Wellcome Trust
Locations (1):
- KEMRI-Wellcome Trust Research Programme, Kilifi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
All trial data will be entered in the clinical trial database, which are maintained through Standard Operating Procedures.
  The volunteer will be identified by a unique trial specific number and/or code in any database. The name and any other identifying detail will NOT be included in any trial data electronic file.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: during study and storage for 10 years
Access Criteria: Direct access will be granted to authorised representatives from the Sponsor, host institution and the regulatory authorities to permit trial-related monitoring, audits and inspections.